CLINICAL TRIAL: NCT01499563
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Antipsychotic Efficacy of ITI-007 in Patients With Schizophrenia
Brief Title: Study of a Novel Antipsychotic ITI-007 in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-005
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ITI-007 Low Dose (Experimental): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered for 28 days
  Interventions: Drug: ITI-007; Drug: Placebo
- ITI-007 High Dose (Experimental): Lumateperone 84 mg (ITI-007 120 mg tosylate) administered for 28 days
  Interventions: Drug: ITI-007
- Placebo (Placebo Comparator): Placebo: Capsules containing inactive placebo administered for 28 days
  Interventions: Drug: Placebo
- Risperidone (Active Comparator): Risperidone: Capsules containing 4 mg risperidone administered for 28 days
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: ITI-007 — Capsules containing ITI-007 for 28 days
  Arms: ITI-007 High Dose; ITI-007 Low Dose
Drug: Placebo — Capsules containing inactive placebo for 28 days
  Arms: ITI-007 Low Dose; Placebo
Drug: Risperidone — Capsules containing risperidone for 28 days
  Arms: Risperidone

SUMMARY:
The purpose of this study is to evaluate whether ITI-007 is effective in reducing symptoms associated with schizophrenia in patients who are having an acute worsening of their psychosis. Patients will be randomly assigned to receive one of two doses of ITI-007, placebo, or a positive control. The primary goal will be to assess the effects of ITI-007 on psychosis. The safety of ITI-007 will also be assessed.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, double-blind, placebo-controlled, multi-center study in patients diagnosed with schizophrenia and an acute exacerbation of psychosis. The efficacy and safety of two dose levels of ITI-007 administered daily for 28 days will be evaluated as compared to placebo; risperidone has been included as a positive control.

Upon completion of the inpatient 28-day Study Treatment Period, patients will be started on standard antipsychotic medication and will be stabilized over a 5-day period before discharge from the study clinic. Patients will be seen for a final outpatient safety evaluation at the End-of-Study visit approximately 2 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is 18-55
* Patient has current diagnosis of schizophrenia and is experiencing an acute exacerbation of psychosis
* Patient has a history of at least three months exposure to one or more antipsychotic therapy(ies) and a prior response to antipsychotic therapy within the previous five years

Exclusion Criteria:

* Any female patient who is pregnant or breast-feeding
* Any patient presenting with concurrent dementia, delirium, mental retardation, epilepsy, drug-induced psychosis, or history of significant brain trauma
* Any patient presenting with schizoaffective disorder, bipolar disorder, acute mania, or major depression with psychotic features
* Any patient considered to be an imminent danger to themselves or others
* Any patient with hematological, renal, hepatic, endocrinological, neurological, or cardiovascular disease or substance abuse as defined by protocol
* Any patient judged by the Investigator to be inappropriate for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly E Vanover, PhD, Study Director — Intra-Cellular Therapies
Locations (8):
- United States (8):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Garden Grove, California
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Rockville, Maryland
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Willingboro, New Jersey
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Austin, Texas

REFERENCES:
- [Derived] Citrome L, Durgam S, Edwards JB, Davis RE. Lumateperone for the Treatment of Schizophrenia: Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. J Clin Psychiatry. 2023 Mar 6;84(2):22r14631. doi: 10.4088/JCP.22r14631. PMID 36883881
- [Derived] Lieberman JA, Davis RE, Correll CU, Goff DC, Kane JM, Tamminga CA, Mates S, Vanover KE. ITI-007 for the Treatment of Schizophrenia: A 4-Week Randomized, Double-Blind, Controlled Trial. Biol Psychiatry. 2016 Jun 15;79(12):952-61. doi: 10.1016/j.biopsych.2015.08.026. Epub 2015 Aug 31. PMID 26444072

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered for 28 days
- Lumateperone 84 mg (ITI-007 120 mg Tosylate): Lumateperone 84 mg (ITI-007 120 mg tosylate) administered for 28 days
- Risperidone 4 mg: Risperidone: Capsules containing 4 mg risperidone administered for 28 days
Period: Overall Study
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
Started | 84 | 83 (84 patients were randomized but only 83 patients received study drug. The number completed and discontinued is based on the 83 patients that received study drug.) | 85 | 82
Completed | 60 | 64 | 61 | 63
Not Completed | 24 | 19 | 24 | 19
Not completed — Withdrawal by Subject | 10 | 11 | 7 | 8
Not completed — Physician Decision | 2 | 1 | 3 | 0
Not completed — Specific Request of Sponsor or Investigator | 2 | 0 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 1 | 6 | 3
Not completed — Other | 8 | 6 | 6 | 4

BASELINE CHARACTERISTICS:
Population: All Baseline data are presented for patients who received at least one dose of study drug, with the exception of the PANSS total score which is presented for patients who received at least 4 doses of study drug and who had a baseline measurement as well as at least 1 valid post-baseline efficacy measurement.
Groups:
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered for 28 days
  Lumateperone 42
- Lumateperone 84 mg (ITI-007 120 mg Tosylate): Lumateperone 84 mg (ITI-007 120 mg tosylate) administered for 28 days
  Lumateperone 84
- Total: Total of all reporting groups
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg | Total
Number analyzed (Participants) | 84 | 83 | 85 | 82 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.03) | 41.4 (8.92) | 40.5 (9.83) | 40.7 (9.33) | 40.1 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 20 | 9 | 58
  Male | 66 | 72 | 65 | 73 | 276
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 13 | 16 | 17 | 16 | 62
  Black or African American | 70 | 62 | 65 | 64 | 261
  Asian | 0 | 0 | 1 | 2 | 3
  Other | 1 | 5 | 3 | 0 | 9
Positive and Negative Syndrome Scale (PANSS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms. Population: PANSS total score Baseline presented for patients who received at least 4 doses of study drug and who had a baseline measurement as well as at least 1 valid post-baseline efficacy measurement (i.e., a measurement after at least 4 doses of study drug).
  units on a scale
    number analyzed (Participants) | 76 | 80 | 80 | 75 | 311
    (all) | 88.1 (11.04) | 84.6 (11.63) | 86.3 (13.10) | 86.1 (12.24) | 86.2 (12.04)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 28 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient, with a score of 1 indicating the absence of symptoms and a score of 7 indicating extremely severe symptoms. Thus, the PANSS Total score minimum is 30 and the maximum is 210, with higher numbers indicating more severe symptoms.
Time Frame: Change from baseline to Day 28
Population: The study was powered for prespecified comparison of both doses of ITI-007 with placebo using a Bonferroni correction for multiple comparisons. The study was not statistically powered to include multiple comparisons of risperidone to placebo and thus, the risperidone 4mg treatment group was included in the model fitting but was not included in the adjustment for multiplicity or primary outcomes determination.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
Number analyzed (Participants) | 76 | 80 | 80 | 75
score on a scale | -13.2 (1.7) | -8.3 (1.7) | -7.4 (1.7) | -13.4 (1.7)
Statistical Analysis 1: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; The study was powered for prespecified comparison of both doses of ITI-007 with placebo using a Bonferroni correction for multiple comparisons. The study was not statistically powered to include multiple comparisons of risperidone to placebo and thus, this comparison is not presented here; Test type: Superiority; p = 0.017, Mixed Effects model for Repeated Measure; Least Squares Mean Difference = -5.8, 95% CI 2-sided [-11.1 to -0.4], Standard Error of Mean 2.4 — 95% CI for LS Mean difference are with Bonferroni correction
Statistical Analysis 2: Comparison: Lumateperone 84 mg (ITI-007 120 mg Tosylate) vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.708, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-6.3 to 4.5], Standard Error of Mean 2.4 — 95% CI for LS Mean difference are with Bonferroni correction

2. Secondary Outcome: Change From Baseline to Day 8 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: as for outcome 1
Time Frame: Change from Baseline to Day 8
Population: ITT Population with LOCF
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
Number analyzed (Participants) | 76 | 80 | 80 | 75
units on a scale | -4.0 (1.2) | -4.7 (1.2) | -2.6 (1.2) | -6.3 (1.2)

3. Secondary Outcome: Change From Baseline to Day 15 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: as for outcome 1
Time Frame: Change from Baseline to Day 15
Population: ITT Population with LOCF
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
Number analyzed (Participants) | 76 | 80 | 80 | 75
units on a scale | -7.8 (1.4) | -4.2 (1.3) | -4.5 (1.3) | -9.6 (1.4)

4. Secondary Outcome: Change From Baseline to Day 22 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: as for outcome 1
Time Frame: Change from Baseline to Day 22
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
Number analyzed (Participants) | 76 | 80 | 80 | 75
units on a scale | -10.5 (1.6) | -6.6 (1.5) | -4.6 (1.5) | -10.8 (1.6)

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~ weeks) including 28 days of double-blind treatment.
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) | Placebo | Risperidone 4 mg
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/83 | 0/85 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83 | 1/85 | 1/82
Other Adverse Events (participants affected / at risk) | 39/84 | 52/83 | 28/85 | 37/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=84) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) (N=83) | Placebo (N=85) | Risperidone 4 mg (N=82)
Psychotic disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=84) | Lumateperone 84 mg (ITI-007 120 mg Tosylate) (N=83) | Placebo (N=85) | Risperidone 4 mg (N=82)
Sedation (Nervous system disorders) | 6 | 17 | 6 | 5
Headache (Nervous system disorders) | 17 | 15 | 11 | 7
Somnolence (Nervous system disorders) | 8 | 11 | 5 | 12
Dizziness (Nervous system disorders) | 5 | 8 | 1 | 1
Akathisia (Nervous system disorders) | 1 | 2 | 2 | 6
Nausea (Gastrointestinal disorders) | 6 | 8 | 1 | 4
Dry Mouth (Gastrointestinal disorders) | 4 | 8 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 1 | 3
Weight Increased (Investigations) | 5 | 5 | 6 | 5
Blood Creatine Phosphokinase Increased (Investigations) | 7 | 3 | 1 | 8
Alanine Aminotransferase Increased (Investigations) | 5 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes